CLINICAL TRIAL: NCT01359540
Title: A Dual Energy X-Ray Absorptiometry (DXA) Evaluation Of Bone Density Changes After Hip Replacement. Performance Of The OMNI Apex Modular™ Hip Stem And The OMNI Apex ARC™ Hip Stem In Primary Total Hip Arthroplasty, Five-Year Clinical And DXA Analysis
Brief Title: Femoral Remodeling Following Total Hip Arthroplasty With OMNI Apex Modular™ and OMNI Apex ARC™ Stem Compared to Competitive Designs
Status: Completed | Type: Observational
Sponsor: Spokane Joint Replacement Center (Other)
Responsible Party: Principal Investigator, David F. Scott, MD, Principle Investigator, Spokane Joint Replacement Center
Other Study IDs: SJRC-OMNH
Record Dates: First submitted 2011-05-22; First posted 2011-05-24 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Osteoarthritis, Hip
Keywords: Total Hip Arthroplasty; Bone Loss; Femoral Remodeling; Bone mineral density; THA; DXA; DEXA; Dual Energy X-Ray Absorptiometry
MeSH Terms: conditions — Osteoarthritis, Hip; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- APEX Modular: APEX Modular Stem group
  Interventions: Device: OMNI Apex Modular™ Hip Device
- ARC Stem: ARC Stem group
  Interventions: Device: OMNI Apex ARC™ Hip Device

INTERVENTIONS:
Device: OMNI Apex Modular™ Hip Device
  Groups: APEX Modular
Device: OMNI Apex ARC™ Hip Device
  Groups: ARC Stem

SUMMARY:
This study compares the change in bone density which occurs after hip replacement with different femoral stem devices.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 20 years, maximum age 80 years
* Osteoarthritis of the hip
* Elective THA
* Signed Informed Consent

Exclusion Criteria:

* Osteoporosis
* Revisions
* Clinically obese (>40 body mass index [BMI])
* Femoral dysplasia
* Trochanteric osteotomy
* Inflammatory arthritis
* Breast-feeding, pregnancy, or women of childbearing potential without documentation of a negative pregnancy test and not utilizing contraception
* Patients with a history of having taken or currently taking bisphosphonates, PTH, fluoride therapy or strontium ranelate or patients taking other chronic medications that in the investigator's opinion are known to affect bone mineral density in a substantial way
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of other investigational agent in the last 30 days
* Unable to sign Informed Consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Femoral bone mineral density | Baseline, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Change in bone mineral density (BMD) as measured by DXA imaging.

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | Pre-operative, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Hip functional outcomes will be assessed using the Harris Hip Score.

CONTACTS AND LOCATIONS:
Overall Officials: David F Scott, MD, Principal Investigator — Spokane Joint Replacement Center
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States